CLINICAL TRIAL: NCT04616456
Title: Effect of Verdiperstat on Microglial Activation in Well-characterized MSA Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Vikram Khurana, MD PhD, Assistant Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003415
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Multiple System Atrophy; Multiple System Atrophy, Cerebellar Variant; Multiple System Atrophy, Parkinson Variant (Disorder); Multiple System Atrophy (MSA) With Orthostatic Hypotension
MeSH Terms: conditions — Multiple System Atrophy; Multiple system atrophy (MSA) with orthostatic hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple System Atrophy (MSA) (Experimental): Twenty to twenty-five subjects with probable MSA diagnosis will be recruited for this study. Each subject will undergo an [F-18]PBR06 PET and MRI scan at baseline, and will receive the experimental drug, verdiperstat (BHV-3241) under supervision of clinic staff. A follow-up [F-18]PBR06 PET and MRI scan will be performed after 6 months (26 weeks) of taking verdiperstat.
  Interventions: Drug: [F-18]PBR06; Drug: Verdiperstat

INTERVENTIONS:
Drug: [F-18]PBR06 — PET radiopharmaceutical
  Other Names: [18-F]PBR06
Drug: Verdiperstat — verdiperstat targets microglial inflammation in the brain
  Other Names: BHV-3241

SUMMARY:
This study will comprise of two phases, an observational phase and a treatment phase.

In the observational phase the specific aims are: 1. To determine the presence and regional distribution of microglial activation, as assessed by 18F-PBR06 PET, in subjects with MSA as compared to healthy controls, at baseline and at 6-9 months' follow-up.

2. To assess the relationship between microglial activation and clinical progression at baseline and follow-up.

In the treatment phase the specific aims of the study are:

The specific aims of the study are:

1. To assess whether verdiperstat (BHV-3241) reduces 18F-PBR06 PET signal, and thus microglial activation and inflammation, in well-characterized MSA patients.
2. To assess the relationship between PET changes and clinical progression at baseline and follow-up in patients treated with verdiperstat.
3. To assess the relationship between PET changes and volumetric brain MRI at baseline and follow-up in patients treated with verdiperstat.

Currently there is no known disease modifying therapy for MSA. Recently, the drug verdiperstat (BHV-3241) has appeared in the investigational arena specifically for the indication of Multiple System Atrophy. Verdiperstat (BHV-3241) is currently being used in a phase 3 active drug trial at Massachusetts Hospital. Verdiperstat (BHV-3241) is known to target Myeloperoxidase, an enzyme implicated in neuroinflammation, a major driver in disease pathogenesis. Our previous study (IRB protocol #2016P002373) demonstrated that applying TSPO (translator protein) PET imaging enabled us to track changes in neuroinflammation and thus provide a viable biomarker for disease progression.

In this pilot study, the investigators aim to assess the effect of an investigational drug, verdiperstat (BHV-3241) on microglial activation in MSA patients using [F-18]PBR06 and to link it with clinical and morphometric MRI brain changes following treatment.

DETAILED DESCRIPTION:
The investigators propose to use a novel TSPO PET ligand, 18F-PBR06 ((18)F-N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline), to assess microglial activation in MSA subjects in response to treatment with verdiperstat.16 [F-18]PBR06 is an arlyoxyanilide-based, second generation TSPO PET ligand that has been demonstrated to have >90% specific binding to their TSPO target in monkey brain.11 It has already been used in humans in dosimetry studies17 and for studies assessing its pharmacokinetic and imaging characteristics in humans16 but has never before been used in MSA subjects until our previous study, IRB protocol #2016P002373. This study will provide a unique opportunity to assess the utility of a novel TSPO PET ligand that has a longer radioisotope half life (approximately, 110 minutes) and hence, has the potential for widespread use depending upon the results of this study. Assessing clinical response in chronic neurodegenerative diseases can be challenging and objective biomarkers are urgently needed. This study would provide pilot data to inform future potential studies using [F-18]PBR06-PET for assessing prognostication, treatment response and drug development for MSA subjects.The investigators intend to recruit MSA patients, one subset for whom the investigators know the longitudinal trajectory of microglial activation changes because of prior participation in IRB protocol # 2016P002373. This will allow us to compare the effects of verdiperstat (BHV-3241) in a well characterized population with each patient serving as his/her own control. To be clear, patients who were not a part of the IRB protocol #2016P002373 will also be offered the study.

The investigators intend to recruit MSA patients in whom the longitudinal trajectory of microglial activation changes has already been determined in IRB protocol # 2016P002373. This will allow us to compare the effects of verdiperstat (BHV-3241) in a well characterized population with each patient serving as his/her own control. However, patients who were not a part of the IRB protocol #2016P002373 will also be offered the study.

The investigators will recruit 8 MSA subjects with previously completed [F-18]PBR06 PET imaging (for protocol #2016P002373) to participate in the study.

The investigators intend to include patients with probable MSA as defined by the following criteria:

* Autonomic failure involving urinary incontinence (inability to control the release of urine form the bladder, with erectile dysfunction in males) or an orthostatic decrease of blood pressure within 3 min of standing by at least 30 mmHg systolic or 15 mm Hg diastolic and
* Poorly levodopa-responsive Parkinsonism (bradykinesia with rigidity, tremor, or postural instability) or
* A cerebellar syndrome (gait ataxia with cerebellar dysarthria, limb ataxia, or cerebellar oculomotor dysfunction) Subjects will be recruited during routine clinical appointments by their physician or one of the other co-investigators listed on the protocol at the Movement Disorders Clinic, 60 Fenwood Road, Boston, MA. All established MSA patients of the Movement Disorders Clinic will be sent a letter describing the study and a copy of the consent form.

ELIGIBILITY:
**Subjects must be located in close proximity to Brigham and Women's Hospital, Boston, MA in order to meet monitoring criteria outlined in study protocol.**

Inclusion/Exclusion criteria:

Subject Inclusion Criteria:

1. Probable MSA clinical diagnosis

Subject Exclusion Criteria:

1. Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
2. Individuals with bipolar disease, schizophrenia, psychotic disorder, or any severe psychiatric disorder
3. History of substance abuse disorder
4. Concurrent medical conditions that contraindicate study procedures
5. Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
6. Individuals with claustrophobia
7. Non-MRI compatible implanted devices
8. Individuals with a genotype indicating that they are low affinity binders of TSPO
9. Abnormal thyroid function (contingent upon free T3, free T4, and TSH levels <10 mIU/L)
10. Renal impairment (RI)
11. Hepatic impairment (HI)
12. Systemic corticosteroid treatment in the past four weeks (excluding nasal or local treatment)
13. Individuals with significant cognitive impairment (i.e. MoCA score less than or equal to 20)
14. Brain MRI indicative of significant abnormality (i.e. prior hemorrhage or infarct)
15. Significant cardiac events within the past year (i.e. hospitalization for congestive heart failure, myocardial infarction, or arrhythmias requiring treatment).
16. Medical conditions that interfere with absorption or secretion of drugs (i.e. gastrointestinal disease)
17. Individuals diagnosed with Human Immunodeficiency Virus Infection Diagnosis (HIV +)
18. Any other clinically significant diagnosis that is currently unstable
19. Hematologic or solid malignancy diagnosis within the past 5 years
20. Medical procedure or surgery within four weeks prior to screening
21. Current treatment through use of any other investigational agent, dopamine antagonists, CYP1A2 inhibitors or inducers, CYP3A4 inhibitors or inducers, or CYP2B6 or CYP3A4 metabolized drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
standardized uptake values (SUV) | 1 month
  PET imaging measurement calculated over whole brain within putamen, pons, cerebellum
standardized uptake ratios (SUVRs) | 1 month
  PET imaging measurement calculated over whole brain within putamen, pons, cerebellum

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Khurana, MD, PhD, Principal Investigator — Brigham and Women's Hospital; Tarun Singhal, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- Movement Disorders Clinic, 60 Fenwood Road, Boston, Massachusetts, United States